CLINICAL TRIAL: NCT04131998
Title: Develop and Validation of Pain Assessment Tools, Back Pain Disability and Autonomy Questionnaires in Albanian Language
Brief Title: Albanian Versions and Validations of Pain Assessment Tools, Back Pain and Autonomy Questionnaires
Acronym: Validation
Status: Completed | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jasemin Todri, Principal Investigator, Universidad Católica San Antonio de Murcia
Other Study IDs: 147/35
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Back Pain; Pain; Disability Physical
MeSH Terms: conditions — Back Pain; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A total of 200 participants are predicted to be enrolled for completing questionnaires in relation of pain assessment tools, back pain disability and autonomy in Albania. A feasibility, validate and test-retest reliability design is estimated.

DETAILED DESCRIPTION:
This study consist of two parts, firstly translation and cross-cultural adaptation of pain and automaton questionnaires into albanian language and secondly psychometric evaluation of the questionnaires including test-retest reliability in Albanian health care centers/ hospitals .

ELIGIBILITY:
Inclusion Criteria:

* back pain
* orthopedic problems
* Albanian citizens
* rehabilitation center patients

Exclusion Criteria:

* neurological patients
* no native albanian language

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Albanian citizens with back pain and with autonomy problems who follows rehabilitation sessions in a rehabilitation center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Pain Assessment Tools | 7 days
  Validation and test-retest of Pain Assessment tools Albanian language. VAS scale consists in identifying the patient, on a 100 cm line, referring to the point that best represents his pain, where 0 means no pain and 100 = worst possible pain.
Roland-Morris Questionnaire (RMQ) for athletes physical disability | 7 days
  Validation of Roland Morrison Questionaire in Albanian language which measures the physical disability of athletes and consists of 24 points of functional capacity of the back. The sense of progression is: the more serious the worse is the performance.
Barthel Index (BI) of patients autonomy | 7 days
  Validation of Barthel Index (BI) in Albanian language. It is used to measure performance in the basic activities of daily life. It refers to the patient's independence in all basic daily living activities. The maximum score used is 100 points and indicates independence in all the basic activities of daily life.
Oswestry Disability Index | 7 days
  Validation o the Oswestry Disability Index in Albanian language is a questionnaire made up of 10 categories: (1) pain intensity, (2) personal care, (3) lifting, (4) walking, (5) sitting, (6) standing, (7) sleeping, (8) sex life, (9) social life, and (10) traveling. Each category consists of 6 items scored from 0 to 5 with the first statement scoring 0 to the last statement scoring 5. A check at the highest levels means the person is in the worst state. If more than one answer is selected, the highest score is considered.

CONTACTS AND LOCATIONS:
Overall Officials: Jasemin Todri, PhD, Principal Investigator — UCAM Universidad Catolica de Murcia
Locations (1):
- Orges Lena, Murcia, España, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Todri J, Gjini E, Lena O. Assessment properties of the Visual Analogue scale, Numeric Rating Scale, Face Pain Scale, and Pain Intensity Subscale of the Brief Pain Inventory in Albanian population with low back pain. Ann Med. 2025 Dec;57(1):2601406. doi: 10.1080/07853890.2025.2601406. Epub 2025 Dec 13. PMID 41388783
- [Derived] Lena O, Todri J. A cross-cultural adaptation study on the validity and test-retest reliability of pain assessment tools in Albanian older adults with low back pain. Geriatr Nurs. 2026 Jan;67:103723. doi: 10.1016/j.gerinurse.2025.103723. Epub 2025 Nov 13. PMID 41237578